CLINICAL TRIAL: NCT06764719
Title: Characterization of Cryopreserved Plucked Hair Follicles and Generation of Functional Cell Lines for Disease Modeling and Cell Replacement Therapies
Brief Title: Cryopreserved Hair Follicles for Disease and Cell Replacement
Status: Recruiting | Type: Observational
Sponsor: Acorn Biolabs Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-003; Company Sponsored (Other: Acorn Biolabs)
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus; Sport Injury; Injury Traumatic
Keywords: Hair follicles; stem cells; pluripotent; cell differentiation
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — hair follicles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hair Follicle Donors: Healthy individuals, aged 18-80, who will have hair follicles collected

SUMMARY:
To explore the application of cells expanded from plucked hair follicles after collection, transport, and cryopreservation, in disease modeling and cell-based therapies.

DETAILED DESCRIPTION:
Hair Follicles collected and transported in Acorn's proprietary transport media can serve has therapeutic starting materials for future cell-based therapeutics. This study is to characterize primary cell outgrowth, functional stem cell generation and induced pluripotent stem cell line(s) from primary outgrowth(s) as well as evaluate and characterize differentiation of stem cell lines into functional cell types required for various disease states and cell-based application(s).

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or Female.
* Age: ≥18 and ≤80 years.
* Language proficiency: Able to read and understand English.
* Informed consent: Willing to provide written, informed consent to participate in all study activities.

Exclusion Criteria:

* Scalp/Hair Disorders: Subjects diagnosed with active scalp infections or inflammatory skin conditions.
* Systemic Conditions: Subjects with chronic illnesses, such as autoimmune diseases or diabetes, that may impact scalp health or wound healing.
* Medications: Subjects on immunosuppressants, steroids, or other medications associated with hair loss.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population, aged 18-80, without scalp or hair disorders, chronic illnesses that may impact scalp health or wound healing, and not on immunosuppressants, steroids, or medications that cause hair loss.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Characterize primary cellular outgrowth(s) | 30 days
  10 hair follicles will be placed in a tissue culture plate per participants. Over the course of 30 days, the outgrowth percentage (the number of outgrowths present out of 10 will be monitored and the confluency (percent of cells present in relation to surface area) will be noted for each participant.
Evaluate functional stem cell generation and induced pluripotent stem cell line(s) from primary outgrowth(s) | 21 days
  1 million keratinocytes will be taken for reprogramming for each participant. The number of iPS colonies observed on day 21 will be noted, resulting in a reprogramming efficiency score.
Evaluate and characterize differentiation of stem cell lines into functional cell types required for various disease states and cell-based application(s) | 30 days
  iPS cell lines which have been confirmed to be pluripotent will be differentiated into pancreatic progenitor cells and hematopoietic stem cells. The cells will be analyzed using FLOW cytometry and the percentage of double positive cells will be noted for each participant. This will be repeated for multiple pathways such as the hematopoietic and endothelial lineage(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Acorn Biolabs, Toronto, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No